

## **DeTACT-AFRICA**

### STATISTICAL ANALYSIS PLAN

A multi-centre randomised controlled non-inferiority trial to compare the efficacy, safety and tolerability of Triple Artemisinin-based Combination Therapies versus first-line ACTs + Placebo for the treatment of uncomplicated Plasmodium falciparum malaria in Africa

A study by the Development of Triple Artemisinin Combination Therapies (DeTACT) Collaboration.

### NCT03923725

ACRONYM: DeTACT Africa study

Version 0.4

Date 16<sup>th</sup> February 2024

| WRITTEN BY: MAVUTO MUKAKA AND CHIRAPORN TAYA | |
|----------------------------------------------|-------|
| PRINT NAME | DATE: |
| STATISTICIAN | |



| REVIEWED AND APPROVED BY: | |
|------------------------------------------|-------|
| DR. MEHUL DHORDA, DR. CHANAKI AMARATUNGA | |
| | DATE: |
| PRINT NAME | |
| PROJECT COORDINATOR | |
| PROF. A.M. DONDORP | |
| | DATE: |
| PRINT NAME | |
| PRINCIPAL INVESTIGATOR | |



# STATISTICAL ANALYSIS PLAN Table of Contents

| <br> | Contonio |
|------|---------------------------|
| 1. | Analysis Considerations |
| 1.1 | General Analysis Approach |

| 1. Analysis Considerations | |
|---|---|
| 1.1 General Analysis Approach | 5 |
| 1.2 Data cleaning and verification | 5 |
| 1.3 Locking the dataset | 5 |
| 1.4 Data format and Analysis logs | 6 |
| 1.5 Interim analyses | 6 |
| 2. Introduction | 6 |
| 2.1. Study objectives and endpoints | 7 |
| 2.1.1. Primary objective | 7 |
| 2.1.2. Primary endpoint | |
| 2.1.3. Secondary objectives and endpoints | 7 |
| 2.1.4. Exploratory objectives and endpoints | 8 |
| 2.2. Study design | |
| 22.1 Determination of sample size | |
| 3. Data Analysis | |
| 3.1 Trial Profile | |
| 3.2 Demographics and other baseline characteristics | |
| 3.3 Efficacy of the ACTs and TACTs as defined by the 42-day PCR corrected adequate clinical and parasitological respon | |
| (ACPR) within each individual site | |
| 3.4 Safety and tolerability of ACTs and TACTs within and across sites and regions, including comparisons of 'non-matchi | |
| ACTs vs TACTs (AL+Placebo versus ASMQ+PPQ, ASMQ+Placebo versus AL+AQ) | 35 |
| 3.5 Changes in the electrocardiogram (such as prolongation of the QTc-interval) in patients treated with TACT versus | |
| standard ACT | |
| 3.7 Pharmacokinetic and pharmacodynamic interactions between antimalarials in ACT and TACTs | |
| 3.8 Molecular genetic and transcriptomic correlates for artemisinin and partner drug resistance of the infecting P. falciparu | |
| strains and to assess their ex vivo and in vitro drug susceptibility | |
| 3.9 In vitro sensitivity of P. falciparum to artemisinins and partner drugs according to study sites and genotype | |
| 3.10 The selective effect of ACTs versus TACTs on parasites carrying mutations associated with resistance to antimalarial | |
| drugs 41 | 40 |
| 3.11 | |
| Change in hematocrit over time according to geographical location and study arm, stratified for G6PD status | |
| 3.12 Correlation between the host genotype (e.g., CYP2D6, CYP3A4, KCNQ1/LQT1, KCNH2/LQT2, SCN5A/LQT3) and the pharmacolkinetics and pharmacolkinetics of antimologicals | |
| pharmacokinetics and pharmacodynamics of antimalarials. | |
| 3.13 Correlations between the place of residence, work, recent travel history assessed by interview and mobile phone recent identify behaviours and risk feeters associated with malaria infection. | |
| to identify behaviours and risk factors associated with malaria infection. | 42 |



| 3.14 Assess new methods for determination of gametocytaemia, parasite phenotypes and genotypes | 42 |
|---|---|
| 3.15 Correlation between specific antibody titres and measures of drug efficacy | . 42 |
| 3.16 Accuracy of SNPs assessment from dry blood spots versus from whole genome sequencing in leukocyte depleted blood | |
| samples | |
| 3.17 Candidate markers of resistance identified through genome wide association studies with in vivo or in vitro parasite drug | |
| | . 42 |
| 3.18 Correlation between qPCR based versus microscopy based assessments of parasite clearance dynamics | . 43 |
| 3.19 Correlation of parasite clearance metrics as assessed by microscopy versus digital microscopy | . 43 |
| 3.20 Comparison of transcriptomic patterns of drug sensitive and resistant parasites before treatment and 6, 12 and 24 hours | |
| after start of treatment | . 43 |
| 3.21 Levels of RNA transcription coding for male or female specific gametocytes at admission up to day 14, stratified by the | |
| presence of gametocytes at enrolment | . 43 |



## 1. Analysis Considerations

#### 1.1 General Analysis Approach

The main analysis strategy for the primary outcome will be the intention-to-treat (ITT) principle. In this analysis, patients will be analysed according to the arm of randomisation irrespective of the treatment that was actually given. Complete Case Analysis will be used in the ITT analysis population (Groenwold et al 2012; Mukaka et al 2016; Sullivan et al 2018). Furthermore, the estimates of efficacy using survival analysis will be done. This approach will help in handling missing data as all patients will be included in the analysis and censored at their last follow-up time. These ITT analyses will be followed by the per protocol (PP) analysis. In this analysis only those that adhered to the protocol with respect to the primary outcome will be included for analysis of the primary outcome.

Key secondary endpoints such as parasite clearance parameters (e.g. half-lives), safety and tolerability data will be analysed similar to the ITT approach for the main primary outcome. In this analysis, patients will be analysed according to the arm of randomisation irrespective of the treatment that was actually given and all patients will be included in the analyses irrespective of their follow-up status as long as they have the data. Withdrawals and losses to follow up will not affect the analyses of this data as long as the relevant data needed for these analyses is available prior to withdrawal or loss to follow up.

Data analysis will mainly be performed using Stata 17 or higher, StataCorp, 4905 Lakeway Drive College Station, Texas 77845 USA or in R software.

## 1.2 Data cleaning and verification

All data will be cleaned and verified prior to statistical analysis. The study site will be visited by the Monitor periodically at times agreed on with the Investigator. At the time of each monitoring visit, the Monitor will review the completed CRFs to ascertain that all items have been completed and that the data provided are accurate and obtained in the manner specified in the protocol. The Monitor will also check that the data in the CRF are consistent with the clinical records (Source Data Verification [SDV]) and that study results are recorded completely and correctly. The data manager will ensure that clean data is submitted to the statistician for analysis. The statistician will cross-check that the available data for analysis is clean. Any data cleaning queries will need to be resolved before statistical analyses.

## 1.3 Locking the dataset

After data cleaning and responding to all data queries, the clean data will be locked normally in the database that was used for data capturing. The data may also be locked and stored in other user-friendly formats such as MS Excel and Stata. The locked data will be stored at an identifiable secure place and should be available to the relevant researchers upon request following proper request procedures.



## 1.4 Data format and Analysis logs

Prior to dispensing data to the trial statistician, the head of data management will make sure that the data to be sent to the trial statistician is clean. This will help the statistician to provide the analysis results in a timely manner as there will be a reduced amount of queries if clean data is provided to the trial statistician. Data will be given to the Trial Statistician by the head of Data Management (or designated person) in a format that is compatible with statistical software reading. Statistical analyses will be performed in Stata, version 17or higher or R software. Statistical programs and output logs will be kept for all analysis and made available upon request.

#### 1.5 Interim analyses

We plan to have 2 interim analyses on clinical, laboratory and electrocardiographic data to assess the safety of the novel TACTs. The interim reports will be reviewed by DSMB. The interim analyses will be performed after the first 100 patients, first 500 patients and at additional time-points before the planned interim analyses, as indicated by the DSMB after their review, if deemed necessary. After this, safety analysis will be performed based on recommendations by the DSMB. No stopping rules both statistical as well as clinical will be specified. The need to stop the trial will be based on the perception of the accumulating data by the DSMB. The main strategy of analysis will focus on safety data although efficacy data may also be presented.

The Trial coordinator in collaboration with the Trial Statistician will produce the report for the DSMB. Only relevant data included in a specific interim report will be made available to the DSMB members at the time of sending the report. During a DSMB meeting, the report will be presented to the members by the study coordinator in line with the meeting agenda. For a normally scheduled DSMB meeting, the report will be sent out to the members at least a week before the meeting.

#### 2. Introduction

This is a multicentre study in 8 different countries in Africa. The study was designed in a way that each centre has 80% power to detect a difference in the efficacy outcomes, if they exist.

Artemisinin combination therapies (ACTs) have been a major contributor to the substantial reductions in global malaria morbidity and mortality over the last decade. However, further gains are threatened by the recent emergence of artemisinin and partner drug resistance in Southeast Asia, a region which has been the epicentre for the evolution and spread of resistance to every important class of antimalarials. Loss of efficacy of first line ACTs jeopardizes current malaria control and elimination efforts and will accelerate the spread of drug resistance. A major concern is that artemisinin and partner drug resistance may spread across a wider geographic area, as chloroquine resistance did in the 1960s and 1970s, moving from Southeast Asia to the Indian subcontinent and subsequently to Africa, which bears the vast majority of the global malaria burden. Furthermore, artemisinin resistance could worsen by extending beyond the current ring stage parasite resistance, although this has until now not been observed. we aim to assess the extent of the spread or the *de novo* emergence of resistance to the antimalarials in the combinations through detailed *in vivo* and *in vitro* assessments and to study the pharmacokinetics and inter-drug interactions of the drugs, the parasite- and host-related factors affecting treatment outcomes. Finally, we aim to gain insights into the spread of resistance mediated by population movements and parasite gene flows in general through travel surveys and geographic localization of parasite genetic data.



The principle that multiple drugs with independent mechanisms of action prevent the emergence of drug resistance is proven in a range of human diseases. In HIV and tuberculosis for example, the occurrence and spread of drug resistance can be prevented by use of a combination of three or more antiretroviral or antimycobacterial therapies respectively, but until now this was not thought necessary in malaria. In malaria there is a fortuitous inverse correlation between susceptibility to artemether-lumefantrine and amodiaquine or artesunate-mefloquine and piperaquine which will be exploited in the TACTs.

### 2.1. Study objectives and endpoints

#### 2.1.1. Primary objective

To compare the efficacy of the ACTs and TACTs as defined by the 42-day PCR corrected adequate clinical and parasitological response (ACPR) within each individual site.

Matching comparisons of ACT and TACT are as follows:

- AL+Placebo versus AL+AQ
- ASMQ+ Placebo versus ASMQ+PPQ

## 2.1.2. Primary endpoint

42-day efficacy defined as PCR-corrected adequate clinical and parasitological response (ACPR).

(NB, WHO definition of ACPR: absence of parasitaemia at day 42 irrespective of axillary temperature and without previously meeting any of the WHO criteria for early or late treatment failure, or late parasitological failure.)

## 2.1.3. Secondary objectives and endpoints

- To compare the safety and tolerability of ACTs and TACTs within and across sites and regions, including comparisons of 'non-matching'
  ACTs vs TACTs (AL+Placebo versus ASMQ+PPQ, ASMQ+Placebo versus AL+AQ).
  - Incidence of adverse events and serious adverse events within the first 42 days including markers of hepatic, renal or bone marrow toxicity; cardiotoxicity, in particular QT or QTc-interval above 500 ms at timepoint H4 and H52/H64 and between these time points; change from baseline in haemoglobin at days 3, 7, 28, stratified for G6PD status/genotype; proportion of subjects requiring retreatment due to vomiting within 1 hour after administration of the study drugs; proportion of subjects that reports completing a full course of observed TACT or ACT without withdrawal of consent or exclusion from study because of drug related serious adverse event
  - Changes in the electrocardiogram (such as prolongation of the QTc-interval) in patients treated with TACT versus standard ACT
- To compare additional measures of treatment efficacy between treatment arms, including the 63-day ACPR, the post-treatment prophylactic
  effect of ACTs and TACTs defined as the 42-day & 63-day PCR uncorrected ACPR, gametocyte carriage, parasite clearance rates and
  fever clearance.



- Comparing 63-day PCR corrected and uncorrected efficacy; 42-day PCR uncorrected efficacy between ACT and TACT
- Parasite clearance half-life assessed by microscopy as primary parameter to determine parasite clearance; proportion of subjects with microscopically detectable P. falciparum parasitaemia at Day 3; fever clearance time (i.e. the time taken for the tympanic temperature to fall below 37.5 °C in patients who were febrile at inclusion); proportion of subjects with gametocytaemia during and after treatment stratified by presence of gametocytes at enrolment.
- To assess pharmacokinetic and pharmacodynamic interactions between antimalarials in ACT and TACTs
  - Pharmacokinetic profiles and interactions (including Cmax and AUC) of artemisinin-derivatives and partner drugs in ACT and TACT treated subjects in correlation with pharmacodynamics measures of drug efficacy; day 7 plasma levels of partner drugs in correlation with treatment efficacy and treatment arm

## 2.1.4. Exploratory objectives and endpoints

- To compare measures of treatment efficacy between treatment arms
  - Comparison of 63-day vs 42-day PCR corrected and uncorrected efficacy of ACTs vs TACTs
- To assess molecular genetic and transcriptomic correlates for artemisinin and partner drug resistance of the infecting *P. falciparum* strains
  - Whole genome sequence and transcriptome analysis of artemisinin and/or partner drug-resistant parasites compared with drugsensitive parasites
- To compare in vitro susceptibility profiles of P. falciparum isolates across geographic regions
  - In vitro sensitivity of P. falciparum to artemisinins and partner drugs according to study sites and genotype
- To compare the selective effect of ACTs versus TACTs on parasites carrying mutations associated with resistance to antimalarial drugs
  - o Proportions of recurrent infections with parasites carrying mutations of known functional significance
  - Proportions of specimens collected at baseline with parasites carrying mutations of known functional or operational significance (pfkelch13, pfcrt, pfmdr1, pfdhfr, pfdhps, pfplasmepsin2, partial or complete deletions of pfhrp2 and other current parasite genetic markers associated with resistance or identified over the course of the study)
- To obtain additional safety data (in particular incidence, rate and magnitude of haemolysis) on the deployment of single low dose primaquine, stratified according to G6PD status/genotype
  - Change in hematocrit on day 1 to 7, 14, 21, 28, 35 and 42 according to geographical location and study arm, stratified for G6PD status
- To obtain additional data on the effect of the host genotypes known to affect pharmacokinetics and pharmacodynamics of antimalarials
  - Correlation between the host genotype (e.g., CYP2D6, CYP3A4, KCNQ1/LQT1, KCNH2/LQT2, SCN5A/LQT3) and the
    pharmacokinetics and pharmacodynamics of antimalarials.
- To assess new methods for determination of gametocytaemia, parasite phenotypes and genotypes
  - Novel assays to be tested



- To assess the correlation between anti-Plasmodium falciparum antibodies and drug efficacy measures
  - Correlation between specific antibody titres and measures of drug efficacy
- To assess and increase the representability/accuracy of parasite genome sequencing from dry blood spots for the genome sequencing results from leukocyte depleted blood samples
  - Accuracy of SNPs assessment from dry blood spots versus from whole genome sequencing in leukocyte depleted blood samples
  - Candidate markers of resistance identified through genome wide association studies with in vitro parasite drug sensitivity phenotypes
  - Correlation between qPCR-based versus microscopy-based assessments of parasite clearance dynamics
  - Correlation of parasite clearance metrics as assessed by microscopy versus digital microscopy
- To identify differences at the transcriptome level in artemisinin and partner drug sensitive and resistant P. falciparum in order to increase
  the understanding of mechanisms of resistance
  - Comparison of transcriptomic patterns of drug sensitive and resistant parasites before treatment and 6, 12 and 24 hours after start of treatment
- To develop DNA and RNA measurement methods for quantification of male and female gametocytes
  - Levels of RNA transcription coding for male or female specific gametocytes at admission up to day 14, stratified by the presence of gametocytes at enrolment

## 2.2. Study design

## **Brief Description**

This is a multi-centre, partially blinded, randomised, controlled non-inferiority trial of the Triple ACTs artemether lumefantrine + amodiaquine (AL+AQ) and artesunate- mefloquine+piperaquine (ASMQ+PPQ)

with the ACTs artemether-lumefantrine + placebo (AL+PBO) and artesunate- mefloquine + placebo (ASMQ+PBO) for the treatment of uncomplicated Plasmodium falciparum malaria to

assess and compare their efficacy, safety, tolerability. The study sites are shown in figure 1 below. Patients will be randomized the ratio 1 ACT: 2:matching TACT to one of the following arms: AL+PBO: AL+AQ: AS-PPQ+MQ: AS-PPQ+PBO.





Figure 1 Study sites

The study will be done in 8 African countries: Burkina Faso, DR Congo, The Gambia, Guinea, Niger, Nigeria, Tanzania and Rwanda.

## 2..2.1 Determination of sample size

These studies will have a non-inferiority trial design. Each site will be powered for the efficacy endpoint. For the safety and tolerability endpoint, the sample size will be pooled across the study sites to achieve the desired power of at least 80% to detect rare events.

For sample size calculations, the following assumptions have been used: The expected efficacy of ACTs (AL, ASMQ) in these countries is expected to be approximately 96%. The matching TACT efficacy is assumed to be at least 90% under the null hypothesis of inferiority based on the WHO 90% efficacy threshold. However preliminary TRACII study data suggest that TACTs potentially may have a better efficacy of 1% to 2% higher in favour of TACT (i.e. a conservative 97%-98% efficacy or higher).

A one-sided alpha of 0.025 has been used in sample size calculations as non-inferiority is in one direction. For the efficacy outcome, a sample size of 60 subjects in the ACT plus placebo arms and 120 subjects in the matching TACT would be needed to achieve approximately 80% power to



detect a non-inferiority margin difference between the group efficacy of -6%. With an additional 20% to cover for loss to follow up, we would therefore need 72 subjects in ACT plus placebo group and 144 subjects in the matching TACT in each of the sites. Since there will be 4 arms, it means we will need 432 subjects per site with 144 subjects in the two ACT arms combined and 288 subjects in the two TACT arms combined.

The sample sizes are in the ratio of 1:2 for ACT vs TACT to allow us to collect more safety and tolerability data for TACTs, which could be beneficial to both policy makers as well as future malaria patients. With these numbers of recruited subjects in Africa, we will have a power above 80% to detect an increase of the incidence of adverse events from 1 in 100 to 3 in 100 for subjects treated with ACT as compared to the matching TACT, respectively.

The sample size calculations were performed using a specialized sample size calculation software, PASS 15.

## 3. Data Analysis

#### 3.1 Trial Profile

The number of patients who will be screened, reasons for non-enrolment, number of patients randomized, number of patients lost to follow up and the number of patients assessed for 42-day endpoint will be summarised in a CONSORT flow diagram, figure 2, below.



#### STATISTICAL ANALYSIS PLAN Assessed for eligibility (N=XXXX) Excluded (N=XXXX) XX Signs of severe/complicated malaria XX Patients not fulfilling criteria for severe malaria but with another indication for parenteral antimalarial treatment at the discretion of the treating physician XX Haematocrit < 15% at screening (<20% for Age of ≥12 years in Gambia site only) XX Subjects who have received artemisinin or a derivative within the previous 7 days OR lumefantrine or amodiaquine within the previous 14 days OR mefloquine or piperaquine within the previous 30 days XX Use of seasonal malaria chemoprophylaxis (SMC) within the last 14 days. XX Acute illness other than malaria requiring systemic treatment XX Severe acute malnutrition (in Niger only) XX Known HIV infection XX Known tuberculosis infection XX For females: post-menarche (in Gambia only) XX History of allergy or known contraindication to any of the study drugs, including neuropsychiatric disorders and epilepsy XX Previous splenectomy XX Enrolment in DeTACT in the previous 3 months XX Participation in another interventional study in the previous 3 months XX Other reasons Enrolled (N=XXXX) and randomised N=XXX assigned and received N=XXX assigned and received AL+AQ N=XXX assigned and received N=XXX assigned and received ASMQ AL+Placebo ASMQ+Placebo +PPQ AL+AQ (N=XXXX) ASMQ +PPQ (N=XXXX) AL+Palcebo (N=XXXX) ASMQ+Placebo (N=XXXX) Safety/ITT analysis Safety/ITT analysis Safety/ITT analysis Safety/ITT analysis XX Study drug discontinued XX Study drug discontinued XX Study drug discontinued XX Study drug discontinued XX Significant non-compliance with XX Significant non-compliance with XX Significant non-compliance with XX Significant non-compliance with treatment treatment regimen treatment regimen treatment regimen reaimen XX An adverse event which requires XX An adverse event which requires XX An adverse event which requires XX An adverse event which requires discontinuation discontinuation discontinuation discontinuation XX Disease progression which XX Disease progression which requires XX Disease progression which requires XX Disease progression which requires requires discontinuation discontinuation discontinuation discontinuation XX Development of severe malaria XX Development of severe malaria XX Development of severe malaria XX Development of severe malaria XX Recurrent parasitaemia XX Recurrent parasitaemia XX Recurrent parasitaemia XX Recurrent parasitaemia XX Loss to follow up XX Loss to follow up XX Loss to follow up XX Loss to follow up ASMQ +PPQ (N=XXXX) AL (N=XXXX) AL+AQ (N=XXXX) ASMQ (N=XXXX) PP analysis PP analysis PP analysis PP analysis

Figure 2 Consort Trial Profile by Arms



## 3.2 Demographics and other baseline characteristics

The following baseline characteristics will be described by study arm in table 1 (below). Variables such as age, heart rate, respiratory rate will be summarized using median and interquartile range (IQR). Continuous variables such as weight, height, systolic and diastolic blood pressure, QT-intervals, haematocrit and haemoglobin will be summarized using mean and standard deviation or median (IQR) as appropriate. Parasitemia at baseline will be described as geometric mean with range. Categorical variables such as sex, presence of fever, bed net use and gametocytemia at baseline will be summarized using frequencies and percentages.

Table 1. Baseline characteristics for the participants per study intervention across the sites

| Characteristics | AL+AQ<br>(N=XX) | AL+Placebo<br>(N=XX) | ASMQ+PP<br>Q<br>(N=XX) | ASMQ+Place<br>bo<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|---|---|
| Female: n (%) | XX(XX.<br>X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Age (years): median (IQR; range) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Age < 12 years: n (%) | XX(XX.<br>X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Pf asexual parasitaemia at hour 0 (/uL): Geometric mean (range)** | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Pf asexual parasitaemia at screening (/uL): Geometric mean (range) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Gametocyte presence; n(%) | XX(XX.<br>X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Haematocrit (%): mean (SD) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X (XX.X) |



| STATISTICAL ANALTSIS FLAN | | | | | |
|---|---|---|---|---|---|
| Weight (kg): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Temperature (°C): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Fever (>=37.5 °C) n (%) | XX(XX.<br>X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Respiratory rate (breaths/min): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Heart rate (beats/min): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Systolic blood pressure (mmHg): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Diastolic blood pressure (mmHg): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Haemoglobin (g/dL): mean (SD) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Creatinine (μMol/L): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| ALT/SGPT (IU/L): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| AST/SGOT(IU/L): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |



| Total Bilirubin (μMol/L): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
|---|---|---|---|---|---|
| Alkaline Phosphatase (IU/L): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| QT interval on monitor (milliseconds): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |
| Calculated QTc Bazett interval (milliseconds): median (IQR) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X<br>(XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) |

## 3.3 Efficacy of the ACTs and TACTs as defined by the 42-day PCR corrected adequate clinical and parasitological response (ACPR) within each individual site

Efficacy will be reported as cumulative ACPR cure rates by day 42 estimated by as day 42 PCR corrected efficacy and compared between ACT vs TACT. The Kaplan Meier/survival methods will be used to visually show time to . Non-inferiority will be assessed using 95% one side confidence intervals.

## Handling of missing data

In the ITT analysis in which efficacy will be reported as proportions of outcomes using Complete case Analysis.

In the PP analysis in which efficacy will be reported as proportions of outcomes, patients in which study drugs are discontinued and/or endpoints are not available due to other reasons (such as withdrawal from the study, loss to follow up, *P falciparum* (Pf) or *P vivax* (Pv) reinfections and inconclusive PCR correction) will be excluded from the analysis.

In the Kaplan-Meier/survival analysis subjects in which study drugs are discontinued and/or endpoints are not available due to other reasons (such as withdrawal from the study, loss to follow up, Pf or Pv reinfections and inconclusive PCR correction) will be censored or treated as competing risks, as appropriate, from the moment of occurrence of one of these events.

Similar analyses as secondary endpoints will be performed for day 63 PCR corrected efficacy and day 42 and day 63 the PCR uncorrected data as well. Where applicable, we will also report the cumulative reinfection rate. The treatment efficacy, 95% confidence intervals and p-values for the comparison of ACTs with matching TACTs will be presented as outlined in tables 2, 3, 4 and 5 below.

Table 2a Comparison of Day 42 PCR corrected Efficacy as proportions of Various ACTs with matching TACTs by sites



| Site | PCR corrected AC n/N, (%) | CPR at day 42, | | Risk difference (95% CI, p-value) | | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Place<br>bo<br>(N=XXXX) | ASMQ + PPQ<br>(N=XXXX) | AL+Placebo vs<br>AL+AQ | ASMQ+Placebo vs<br>ASMQ+PPQ |
| Burkina<br>Faso | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| DR<br>Congo | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Gambia | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Guinea | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Niger | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Nigeria | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Tanzania | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Rwanda | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| All sites | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |







Difference in percentage of Day 42 PCR corrected Efficacy (95% CI)



## Figure 3 The difference between TACT vs ACT of Day 42 PCR corrected Efficacy as proportions by site

Table 2b Comparison of Day 42 PCR corrected Efficacy using survival methods of Various ACTs with matching TACTs by sites

| Site | PCR corrected ACPR Cumulative recurrent in | at day 42,<br>nfection free percentage | e (efficacy), % (95% | CI) | Hazard ratio (95% CI, p-value) | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Placebo<br>(N=XXXX) | ASMQ +<br>PPQ<br>(N=XXXX) | AL+Placebo vs AL+AQ | ASMQ+Placebo<br>vs ASMQ+PPQ |
| Burkina<br>Faso | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| DR<br>Congo | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Gambia | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Guinea | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Niger | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Nigeria | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Tanzania | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Rwanda | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| All sites | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |





Figure 4.1 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in Burkina Faso

Figure 4.2 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in DR Congo

Figure 4.3 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in Gambia

Figure 4.4 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in Guinea



Figure 4.5 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in Niger

Figure 4.6 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in Nigeria

Figure 4.7 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in Tanzania

Figure 4.8 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in Rwanda

Figure 4.9 Cumulative recurent infection free probability until day 42 from PCR corrected by treatment in all sites

Table 3a Comparison of Day 63 PCR corrected Efficacy as proportions of Various ACTs with matching TACTs by sites

| Site | PCR corrected AC n/N, (%) | CPR at day 63, | | Risk difference (95% CI, p-value) | | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Place<br>bo<br>(N=XXXX) | ASMQ + PPQ<br>(N=XXXX) | AL+Placebo vs<br>AL+AQ | ASMQ+Placebo vs<br>ASMQ+PPQ |
| Burkina<br>Faso | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| DR<br>Congo | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Gambia | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Guinea | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Niger | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Nigeria | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Tanzania | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Rwanda | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |



| All sites | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
|---|---|---|---|---|---|---|
| All Siles | | | (XX.X) | | 0.XXX) | |







Difference in percentage of Day 63 PCR corrected Efficacy (95% CI)



## Figure 5 The difference between TACT vs ACT of Day 63 PCR corrected Efficacy as proportions by site

Table 3b Comparison of Day 63 PCR corrected Efficacy using survival methods of Various ACTs with matching TACTs by sites

| Site | PCR corrected ACPR Cumulative recurrent i | at day 63,<br>nfection free percentage | e (efficacy), % (95% | CI) | Hazard ratio (95% CI, p-value) | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Placebo<br>(N=XXXX) | ASMQ +<br>PPQ<br>(N=XXXX) | AL+Placebo vs AL+AQ | ASMQ+Placebo<br>vs ASMQ+PPQ |
| Burkina<br>Faso | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| DR<br>Congo | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Gambia | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Guinea | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Niger | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Nigeria | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Tanzania | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Rwanda | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| All sites | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |





Figure 6.1 Cumulative recurent infection free probability until day 63 from PCR corrected and days by treatment in Burkina Faso

Figure 6.2 Cumulative recurent infection free probability until day 63 from PCR corrected and days by treatment in DR Congo Figure 6.3 Cumulative recurent infection free probability until day 63 from PCR corrected by treatment in Gambia

Figure 6.4 Cumulative recurent infection free probability until day 63 from PCR corrected by treatment in Guinea



Figure 6.5 Cumulative recurent infection free probability until day 63 from PCR corrected by treatment in Niger

Figure 6.6 Cumulative recurent infection free probability until day 63 from PCR corrected by treatment in Nigeria

Figure 6.7 Cumulative recurent infection free probability until day 63 from PCR corrected by treatment in Tanzania

Figure 6.8 Cumulative recurent infection free probability until day 63 from PCR corrected and days by treatment in Rwanda

Figure 6.9 Cumulative recurent infection free probability until day 63 from PCR corrected and days by treatment in all sites

Table 4a Comparison of Day 42 PCR uncorrected Efficacy as proportions of Various ACTs with matching TACTs by sites

| Site | PCR uncorrected n/N, (%) | ACPR at day 42, | | | Risk difference (95% CI, p-value) | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Place<br>bo | ASMQ + PPQ<br>(N=XXXX) | AL+Placebo vs<br>AL+AQ | ASMQ+Placebo vs<br>ASMQ+PPQ |
| Burkina<br>Faso | XX/XXX (XX.X) | XX/XXX (XX.X) | (N=XXXX)<br>XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| DR<br>Congo | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Gambia | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Guinea | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |



| Nigor | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
|---|---|---|---|---|---|---|
| Niger | , , | , , | (XX.X) | , , | 0.XXX) | , , |
| Nigeria | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
| Nigeria | | | (XX.X) | | 0.XXX) | |
| Tanzania | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
| Tarizarila | | | (XX.X) | | 0.XXX) | |
| Rwanda | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
| itwanua | | | (XX.X) | | 0.XXX) | |
| All sites | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
| All Siles | | | (XX.X) | | 0.XXX) | |







Difference in percentage of Day 42 PCR uncorrected Efficacy (95% CI)



## Figure 7 The difference between TACT vs ACT of Day 42 PCR uncorrected Efficacy as proportions by site

Table 4b Comparison of Day 42 PCR uncorrected Efficacy using survival methods of Various ACTs with matching TACTs by sites

| Site | PCR uncorrected ACP Cumulative recurrent in | PR at day 42,<br>nfection free percentage | e (efficacy), % (95% | CI) | Hazard ratio (95% Cl, p-value) | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Placebo<br>(N=XXXX) | ASMQ +<br>PPQ<br>(N=XXXX) | AL+Placebo vs AL+AQ | ASMQ+Placebo<br>vs ASMQ+PPQ |
| Burkina<br>Faso | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| DR<br>Congo | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Gambia | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Guinea | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Niger | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Nigeria | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Tanzania | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Rwanda | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| All sites | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |





Figure 8.1 Cumulative recurent infection free probability until day 42 from PCR uncorrected and days by treatment in Burkina Faso

Figure 8.2 Cumulative recurent infection free probability until day 42 from PCR uncorrected and days by treatment in DRC Congo Figure 8.3 Cumulative recurent infection free probability until day 42 from PCR uncorrected by treatment in Gambia

Figure 8.4 Cumulative recurent infection free probability until day 42 from PCR uncorrected by treatment in Guinea

Figure 8.5 Cumulative recurent infection free probability until day 42 from PCR uncorrected by treatment in Niger



Figure 8.6 Cumulative recurent infection free probability until day 42 from PCR uncorrected by treatment in Nigeria

Figure 8.7 Cumulative recurent infection free probability until day 42 from PCR uncorrected by treatment in Tanzania

Figure 8.8 Cumulative recurent infection free probability until day 42 from PCR uncorrected and days by treatment in Rwanda

Figure 8.9 Cumulative recurent infection free probability until day 42 from PCR uncorrected and days by treatment in all sites

Table 5a Comparison of Day 63 PCR uncorrected Efficacy as proportions of Various ACTs with matching TACTs by sites

| Site | PCR uncorrected n/N, (%) | ACPR at day 63, | | | Risk difference (95% CI, p-value) | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Place<br>bo<br>(N=XXXX) | ASMQ + PPQ<br>(N=XXXX) | AL+Placebo vs<br>AL+AQ | ASMQ+Placebo vs<br>ASMQ+PPQ |
| Burkina<br>Faso | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| DR<br>Congo | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Gambia | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Guinea | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |
| Niger | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX<br>(XX.X) | XX/XXX (XX.X) | XX.X (XX.X - XX.X,<br>0.XXX) | XX.X (XX.X - XX.X, 0.XXX) |



| Nigeria | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
|---|---|---|---|---|---|---|
| ivigeria | | | (XX.X) | | 0.XXX) | |
| Tanzania | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
| Tarizariia | | | (XX.X) | | 0.XXX) | |
| Rwanda | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
| Rwanua | | | (XX.X) | | 0.XXX) | |
| All sites | XX/XXX (XX.X) | XX/XXX (XX.X) | XX/XXX | XX/XXX (XX.X) | XX.X (XX.X - XX.X, | XX.X (XX.X - XX.X, 0.XXX) |
| All Siles | | | (XX.X) | | 0.XXX) | |







Difference in percentage of Day 63 PCR uncorrected Efficacy (95% CI)



## Figure 9 The difference between TACT vs ACT of Day 63 PCR uncorrected Efficacy as proportions by site

## Table 5b Comparison of Day 63 PCR uncorrected Efficacy using survival methods of Various ACTs with matching TACTs by sites

| Site | PCR uncorrected ACF<br>Cumulative recurrent i | PR at day 63,<br>nfection free percentage | e (efficacy), % (95% | CI) | Hazard ratio (95% CI, p-value) | |
|---|---|---|---|---|---|---|
| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Placebo<br>(N=XXXX) | ASMQ +<br>PPQ<br>(N=XXXX) | AL+Placebo vs AL+AQ | ASMQ+Placebo<br>vs ASMQ+PPQ |
| Burkina<br>Faso | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| DR<br>Congo | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Gambia | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Guinea | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Niger | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Nigeria | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Tanzania | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| Rwanda | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |
| All sites | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X -<br>XX.X) | XX.X<br>(XX.X -<br>XX.X) | XX.X (XX.X - XX.X, 0.XXX) | XX.X (XX.X -<br>XX.X, 0.XXX) |





Figure 10.1 Cumulative recurent infection free probability until day 63 from PCR uncorrected and days by treatment in Burkina Faso

Figure 10.2 Cumulative recurent infection free probability until day 63 from PCR uncorrected and days by treatment in DRC Congo Figure 10.3 Cumulative recurent infection free probability until day 63 from PCR uncorrected by treatment in Gambia

Figure 10.4 Cumulative recurent infection free probability until day 63 from PCR uncorrected by treatment in Guinea

Figure 10.5 Cumulative recurent infection free probability until day 63 from PCR uncorrected by treatment in Niger



Figure 10.6 Cumulative recurent infection free probability until day 63 from PCR uncorrected by treatment in Nigeria

Figure 10.7 Cumulative recurent infection free probability until day 63 from PCR uncorrected by treatment in Tanzania

Figure 10.8 Cumulative recurent infection free probability until day 63 from PCR uncorrected and days by treatment in Rwanda

Figure 10.9 Cumulative recurent infection free probability until day 63 from PCR uncorrected and days by treatment in all sites

# 3.4 Safety and tolerability of ACTs and TACTs within and across sites and regions, including comparisons of 'non-matching' ACTs vs TACTs (AL+Placebo versus ASMQ+PPQ, ASMQ+Placebo versus AL+AQ).

Safety analyses will be based on the whole population that get administered the study drug. That is, the safety and tolerability data will be pooled from all the sites that received the same antimalarial treatment. Safety and tolerability of TACTs versus ACTs will be assessed by comparing the frequency (%) of adverse events and serious adverse events, with particular attention to abdominal pain, appetite perturbation, biochemical markers of hepatic and renal toxicity and QT interval prolongation, using the Fisher's exact test. Safety data will be presented in tabular and/or graphical format and summarized descriptively. Any clinically relevant abnormalities or values of potential clinically concern will be described. Patients will be analysed following the intention to treat analysis. All adverse event summaries will refer to treatment emergent adverse events, i.e. adverse events that newly started or increased in intensity after the study drug administration. Adverse events will be graded according to Division of AIDS table for grading the severity of ADULT AND PEDIATRIC adverse Events Version 2.0, November, 2014. The relevant DAIDS table will be appended to this document. The safety and tolerability summaries will be presented in tables 6.

The frequency and proportion of subjects that reports completing a full course of observed TACT or ACT without withdrawal of consent or exclusion from study because of drug related serious adverse events will be summarized within and across sites and regions. The 95% confidence intervals will be reported for the proportions. The proportions will be compared between matching drugs. The analyses will be summarised in table 7.

## 3.5 Changes in the electrocardiogram (such as prolongation of the QTc-interval) in patients treated with TACT versus standard ACT

Incidence of prolongations of the QTc-interval (QTc Bazett)>500 miliseconds at least once (at H4, H48, H52) will be summarized in table 5. Absolute changes in the QTc-interval will be summarized as in tables 8, and will be graphically displayed by arm as in figure 5. Comparisons on the changes in the QTc-interval will be made using the unpaired t-test for each specific time point.



## Table 6 Adverse events within the first 42 days

| Adverse events | AL+Placebo | | AL+AQ | | ASMQ+Pla | icebo | ASMQ + I | PPQ |
|---|---|---|---|---|---|---|---|---|
| Number of subjects | XXXX | | XXXX | | XXXX | | XXXX | |
| Vomiting/number of treatments, n/N, (%) | XXX/> | XXXX (XX.X) | XXX/XXX | X (XX.X) | XXX/XX> | XX (XX.X) | XXX/XXX | X (XX.X) |
| Serious adverse events (SAEs) , n/N, (%) | XX/> | XXXX (XX.X) | XX/XXX | X (XX.X) | XX/XX> | (X (XX.X) | XX/XXX | X (XX.X) |
| Possible, probable or definite drug related SAEs, n/N, (%) | XX/> | XXXX (XX.X) | XX/XXX | X (XX.X) | XX/XX> | (X (XX.X) | XX/XXX | X (XX.X) |
| QTc >500ms (H4 and H48/H52) | XXX/> | XXXX (XX.X) | XXX/XXX | X (XX.X) | XXX/XX> | XX (XX.X) | XXX/XXX | X (XX.X) |
| Change from baseline in haemoglobin at days 3, 7, 28 (stratified for G6PD status) | XXX/X | XXXX (XX.X) | XXX/XXX | X (XX.X) | XXX/XXX | (X (XX.X) | XXX/XXX | X (XX.X) |
| Grading of adverse events, n/N, (%) | 1-2 | 3-4 | 1-2 | 3-4 | 1-2 | 3-4 | 1-2 | 3-4 |
| Symptoms, n/N (%) | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Headache | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Fatigue | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Abdominal pain | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Loss of appetite | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Nausea | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Vomiting | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Diarrhea | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Itching | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Dizziness | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |
| Blurred vision | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) | X/XX<br>(X.X) |



| Sleeping disturbance | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX | X/XX | X/XX | X/XX | X/XX |
|---|---|---|---|---|---|---|---|---|
| | | | | (X.X) | (X.X) | (X.X) | (X.X) | (X.X) |
| Laboratory abnormalities, n/N (%) | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX | X/XX | X/XX | X/XX | X/XX |
| | | | | (X.X) | (X.X) | (X.X) | (X.X) | (X.X) |
| Creatinine | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX | X/XX | X/XX | X/XX | X/XX |
| | | | | (X.X) | (X.X) | (X.X) | (X.X) | (X.X) |
| Total bilirubine | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX | X/XX | X/XX | X/XX | X/XX |
| | | | | (X.X) | (X.X) | (X.X) | (X.X) | (X.X) |
| Alkaline phosphatase | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX | X/XX | X/XX | X/XX | X/XX |
| | | | | (X.X) | (X.X) | (X.X) | (X.X) | (X.X) |
| Alanyl transfarase (ALT) | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX | X/XX | X/XX | X/XX | X/XX |
| | | | | (X.X) | (X.X) | (X.X) | (X.X) | (X.X) |
| Aspartate transfarase (AST) | X/XX (X.X) | X/XX (X.X) | X/XX (X.X) | X/XX | X/XX | X/XX | X/XX | X/XX |
| | | | | (X.X) | (X.X) | (X.X) | (X.X) | (X.X) |

QTc: QT corrected using Bazett's formula. Adverse event grading: grade1: mild; grade 2: moderate; grade 3: severe; grade 4: potentially life-threatening

Incidence of QTc abnormalities (>500 miliseconds) and bradycardia is defined as a subjects experience these abnormalities at one or more timepoints.

Table 7a Proportions of patients that report a full course of observed TACT or ACT

| | AL,<br>n/N (%, 95% CI) | A+AQ,<br>n/N (%, 95% CI) | ASMQ,<br>n/N (%, 95% CI) | ASMQ + PPQ,<br>n/N (%, 95% CI) | p-value<br>(AL vs<br>AL+AQ) | p-value<br>(ASMQ vs<br>ASMQ+PPQ) |
|---|---|---|---|---|---|---|
| Completing full course of study drug | XXXX/XXXX (XX.X,<br>XX.X - XX.X) | XXXX/XXXX (XX.X,<br>XX.X - XX.X) | XXXX/XXXX (XX.X,<br>XX.X - XX.X) | XXXX/XXXX (XX.X,<br>XX.X - XX.X) | 0.XXX | 0.XXX |

Table 7b. Necessity for retreatment due to vomiting or spitting study drug

| | AL+AQ | AL+Placeb<br>o | ASMQ+PP<br>Q | ASMQ+Placebo |
|---|---|---|---|---|
| Number of participants | XX | XX | XX | XX |
| Number of total doses | XX | XX | XX | XX |



| Retreatment events | | | | |
|---|---|---|---|---|
| Number of participants | XX | XX | XX | XX |
| Retreatment events due to vomiting (< 30 min) only† | X(X) | X(X) | X(X) | X(X) |
| Retreatment events due to spitting only† | X(X) | X(X) | X(X) | X(X) |
| Both vomit and spitting*† | X(X) | X(X) | X(X) | X(X) |
| Total number of retreatments† | X(X) | X(X) | X(X) | X(X) |
| Total number of participants vomiting after retreatment (< 60 min) or rescue therapy given | X(X) | X(X) | X(X) | X(X) |
| Number of participants vomiting after retreatment (< 60 min) | X(X) | X(X) | X(X) | X(X) |
| Number of rescue treatments given | X(X) | X(X) | X(X) | X(X) |

Table 8 QTc-intervals and changes in QTcintervals over time (relevant time points only will be summarised)

| Time- | AL+Placebo | | | AL+AQ | | ASMQ+Placebo | | | ASMQ+PPQ | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| point | QTc | Δ-QTc | p-value | QTc | Δ-QTc | p-value | QTc | Δ-QTc | p-value | QTc | Δ-QTc | p-value |
| H0 | XXX.X<br>(XX.X) | Baseline | Baseline | XXX.X<br>(XX.X) | Baseline | Baseline | XXX.X<br>(XX.X) | Baseline | Baseline | XXX.X<br>(XX.X) | Baseline | Baseline |
| H4 | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX |
| H24 | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX |
| H28 | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX |
| H48 | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX | XXX.X<br>(XX.X) | XX.X<br>(XX.X) | 0.XXX |



| H52 | XXX.X | XX.X | 0.XXX | XXX.X | XX.X | 0.XXX | XXX.X | XX.X | 0.XXX | XXX.X | XX.X | 0.XXX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | |
| H60 | XXX.X | XXX.X | 0.XXX | XXX.X | XXX.X | 0.XXX | XXX.X | XXX.X | 0.XXX | XXX.X | XXX.X | 0.XXX |
| | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | |
| H64 | XXX.X | XXX.X | 0.XXX | XXX.X | XXX.X | 0.XXX | XXX.X | XXX.X | 0.XXX | XXX.X | XXX.X | 0.XXX |
| | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | |

# 3.6 Assessing and comparing P. falciparum parasite clearance rate, additional parameters of parasite clearance dynamics and fever clearance time of standard ACTs and matching TACTs.

Parasite clearance half-life, proportion of subjects with microscopically detectable P. falciparum parasitaemia at Day 3 and fever clearance time (i.e. the time taken for the tympanic temperature to fall below 37.5 °C in patients who were febrile at inclusion) will be summarized and presented in table 9 below. In addition, proportion of subjects with gametocytaemia during and after treatment stratified by presence of gametocytes at enrolment will be presented in tables 9 and 10 below.

Table 9. Parasite clearance half-life, microscopy P. falciparum positivity and fever clearance time (up to H72 vs after H72)

| Arms | Median Time (hours) to Resolution of Fever (range) * | Median<br>Parasite<br>Clearance<br>Half-Life in<br>hours (range) | Median Time (hours) to 50% Parasite Clearance (range) ** | Median Time (hours) to 90% Parasite Clearance (range) ** | Parasite<br>Clearance<br>Half-Life >5 hours,<br>(n/N) % (95% CI) ** | Positive<br>for Parasitaemia<br>on day 3, (n/N) %<br>(95% CI) *** |
|---|---|---|---|---|---|---|
| AL based overall | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | (XX/XX) X(X–X) | (XX/XX) X(X–X) |
| AL+AQ | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | (XX/XX) X(X–X) | (XX/XX) X(X–X) |
| AL+Placebo | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | (XX/XX) X(X–X) | (XX/XX) X(X–X) |
| ASMQ based overall | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | (XX/XX) X(X–X) | (XX/XX) X(X–X) |
| ASMQ +PPQ | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | (XX/XX) X(X–X) | (XX/XX) X(X–X) |



| ASMQ | XX.X (XX.X-XX.X) | XX.X (XX.X- | XX.X (XX.X-XX.X) | XX.X (XX.X- | (XX/XX) X(X-X) | (XX/XX) X(X–X) |
|---|---|---|---|---|---|---|
| +Placebo | | XX.X) | | XX.X) | | |

Table 10 Gametocytaemia during and after treatment by gametocytes status at enrolment

| | | p-value<br>(AL+Placebo | p-value<br>(ASMQ+Placebo | | | |
|---|---|---|---|---|---|---|
| | AL+Placebo | AL+AQ | ASMQ+Placebo | ASMQ + PPQ | vs AL+AQ) | vs ASMQ+PPQ) |
| Presence of gametocytes at enrolment | (N=XXXX) | (N=XXXX) | (N=XXXX) | (N=XXXX) | | |
| During treatment | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X,<br>XX.X-XX.X) | 0.XXX | 0.XXX |
| After treatment | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X,<br>XX.X-XX.X) | 0.XXX | 0.XXX |
| Absence of gametocytes at enrolment | (N=XXXX) | (N=XXXX) | (N=XXXX) | (N=XXXX) | | |
| During treatment | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X,<br>XX.X-XX.X) | 0.XXX | 0.XXX |
| After treatment | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X,<br>XX.X-XX.X) | 0.XXX | 0.XXX |

## 3.7 Pharmacokinetic and pharmacodynamic interactions between antimalarials in ACT and TACTs

A detailed analysis plan will be prepared separately.

# 3.8 Molecular genetic and transcriptomic correlates for artemisinin and partner drug resistance of the infecting P. falciparum strains and to assess their ex vivo and in vitro drug susceptibility

A detailed analysis plan will be prepared separately.

## 3.9 In vitro sensitivity of P. falciparum to artemisinins and partner drugs according to study sites and genotype

A detailed analysis plan will be prepared separately.



# 3.10 The selective effect of ACTs versus TACTs on parasites carrying mutations associated with resistance to antimalarial drugs

Recurrent infections with parasites carrying mutations of known functional significance and specimens collected at baseline with parasites carrying mutations of known functional or operational significance (pfkelch13, pfcrt, pfmdr1, pfdhfr, pfdhps, pfplasmepsin2, partial or complete deletions of pfhrp2 and other current parasite genetic markers associated with resistance or identified over the course of the study) will be summarized as proportions of the total number of samples per site (% and 95% confidence interval) as in table 11.

Table 12 Recurrent infections and specimens collected at baseline with parasites carrying mutations of known functional significance

| | AL+Placebo<br>(N=XXXX) | AL+AQ<br>(N=XXXX) | ASMQ+Placebo<br>(N=XXXX) | ASMQ + PPQ<br>(N=XXXX) | p-value<br>(AL+Placebo<br>vs AL+AQ) | p-value<br>(ASMQ+Placebo<br>vs ASMQ+PPQ) |
|---|---|---|---|---|---|---|
| Reinfections, n (%,CI 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Pf kelch13, n (%,Cl 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Pf crt, n (%,CI 95%) | XX (XX.X,<br>XX.X-XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | XX (XX.X, XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Pf mdr1, n (%,Cl 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Pf dhfr, n (%,Cl 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Pf dhps, n (%,Cl 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Pf Plasmepsin 2, n (%,Cl 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Partial or complete<br>deletions of PF hrp2, n<br>(%,CI 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |
| Others, n (%,Cl 95%) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-<br>XX.X) | XX.X (XX.X-<br>XX.X) | 0.XXX | 0.XXX |



3.11

## Change in hematocrit over time according to geographical location and study arm, stratified for G6PD status

Change in hematocrit on day 1 to 7, 14, 21, 28, 35 and 42 according to geographical location and study arm, stratified for G6PD status will be summarized and analyzed. A detailed analysis plan will be prepared separately.

3.12 Correlation between the host genotype (e.g., CYP2D6, CYP3A4, KCNQ1/LQT1, KCNH2/LQT2, SCN5A/LQT3) and the pharmacokinetics and pharmacodynamics of antimalarials.

A detailed analysis plan will be prepared separately.

3.13 Correlations between the place of residence, work, recent travel history assessed by interview and mobile phone records to identify behaviours and risk factors associated with malaria infection.

A detailed analysis plan will be prepared separately.

3.14 Assess new methods for determination of gametocytaemia, parasite phenotypes and genotypes

A detailed analysis plan will be prepared separately.

3.15 Correlation between specific antibody titres and measures of drug efficacy

A detailed analysis plan will be prepared separately.

3.16 Accuracy of SNPs assessment from dry blood spots versus from whole genome sequencing in leukocyte depleted blood samples

A detailed analysis plan will be prepared separately.

3.17 Candidate markers of resistance identified through genome wide association studies with in vivo or in vitro parasite drug sensitivity phenotypes

A detailed analysis plan will be prepared separately.



3.18 Correlation between qPCR based versus microscopy based assessments of parasite clearance dynamics

A detailed analysis plan will be prepared separately.

3.19 Correlation of parasite clearance metrics as assessed by microscopy versus digital microscopy

A detailed analysis plan will be prepared separately.

3.20 Comparison of transcriptomic patterns of drug sensitive and resistant parasites before treatment and 6, 12 and 24 hours after start of treatment

A detailed analysis plan will be prepared separately.

3.21 Levels of RNA transcription coding for male or female specific gametocytes at admission up to day 14, stratified by the presence of gametocytes at enrolment

A detailed analysis plan will be prepared separately.